CLINICAL TRIAL: NCT05438641
Title: Retrospective Chart Review of Treatment of Alcohol Withdrawal Syndrome With Alpha-2 Agonists and/or Anticonvulsants
Brief Title: Treatment of Alcohol Withdrawal Syndrome With Alpha-2 Agonists and/or Anticonvulsants
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 25510
Record Dates: First submitted 2014-04-15; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: Alcohol withdrawal; withdrawal seizures; DT; delirium tremens; rum fits; the shakes
MeSH Terms: conditions — Alcohol Withdrawal Delirium; Alcohol Withdrawal Seizures; Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Benzodiazepine-based treatment group: Conventional Benzodiazepine-based group includes any subject primarily treated with BZDP agents (e.g., diazepam, lorazepam, chlordiazepoxide).
  Interventions: Drug: BZDP-Based Protocol
- Benzodiazepine-Sparing: BZDP-Sparing group includes subjects primarily treated with a non-BZDP agent (e.g., Alpha-2 agonists and/or anticonvulsants).
  Interventions: Drug: BZDP-Sparing Protocol

INTERVENTIONS:
Drug: BZDP-Sparing Protocol — BZDP-Sparing group includes subjects primarily treated with a non-BZDP agent (e.g., Alpha-2 agonists and/or anticonvulsants). Rescue with BZDP-based treatment allowed if there is symptomatic breakthrough- as measured by CIWA > 15.
  Groups: Benzodiazepine-Sparing
Drug: BZDP-Based Protocol — Patients in this arm will received active treatment based on conventional BZDP-based protocol; additional BZDP are permitted for patients who are still symptomatic, based on CIWA-Protocol.
  Other Names: Conventional Treatment
  Groups: Conventional Benzodiazepine-based treatment group

SUMMARY:
Complicated alcohol withdrawal syndrome (AWS) increases morbidity and mortality of hospitalized, medically ill patients. The Psychosomatic Medicine Service is commonly consulted to assist in the management of these patients when admitted to medical/surgical units. During the last 15 months, the investigators have implemented a benzodiazepine-sparing management approach with very positive clinical outcomes. The BZDP-sparing protocol consists of a combination of alpha-2 agonist and/or anticonvulsant agents; all currently being used for the management of other medical conditions. This project intends to collect and analyze the data of all subjects managed with this approach to better understand its effectiveness and assess for potential adverse effects.

DETAILED DESCRIPTION:
Complicated alcohol withdrawal syndrome (C-AWS) increases morbidity and mortality of hospitalized, medically ill patients. The Psychosomatic Medicine Service is commonly consulted to assist in the management of these patients when admitted to medical/surgical units. During the last 15 months, the investigators have implemented a benzodiazepine-sparing management approach with very positive clinical outcomes. The BZDP-sparing protocol consists of a combination of alpha-2 agonist (e.g., clonidine, guanfacine, dexmedetomidine) and/or anticonvulsant agents (e.g., gabapentin, valproic acid, carbamazepine); all currently being used for the management of other medical conditions. The proposed study consists of an exhaustive chart review of these records to better understand the safety and effectiveness of alpha-2 agonists and anticonvulsants in the prophylaxis and treatment of AWS. Specifically the investigators want to understand the time to resolution of AWS symptoms, whether there are any limiting side effects to this regimen, and the need of for rescue with benzodiazepine agents. The information obtained from this study will be very helpful in assisting in the design of safer and more effective treatment of AWS.

ELIGIBILITY:
Inclusion Criteria:

* All the cases referred to the Psychosomatic Medicine Service for assistance with prophylactic or symptomatic management of AWS starting 8/1/2011 until 8/31/2014.

Exclusion Criteria:

* Patients who through chart review were found to have been primarily suffering from delirium from causes other than AWS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be 18 year old and older patients treated at Stanford Hospital for AWS by CL Psychiatry. The subjects will be of both genders and any ethnic background.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Institute Withdrawal Assessment for Alcohol (CIWA) Score | Baseline to month 6
  The Clinical Institute Withdrawal Assessment for Alcohol (CIWA) measure is a ten item measure of alcohol withdrawal symptoms. The CIWA total score is the summation of 10 questions, with a range from 0 (little to no withdrawal) to 67 (worse alcohol withdrawal).

SECONDARY OUTCOMES:
Treatment Safety | Up to 6 months
  Presence and nature of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maldonado, MD, Principal Investigator — Stanford University Department of Psychiatry
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States